CLINICAL TRIAL: NCT02752568
Title: Assisted Hatching Versus Endometrial Scratch in Recurrent Implantation Failure.A Comparative Study
Brief Title: Assisted Hatching Versus Endometrial Scratch in Recurrent Implantation Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, suzy abdelaziz Abdelhamid, lecturer of obstetrics & gynecology, Kasr El Aini Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: ivfobgyn
Record Dates: First submitted 2016-04-25; First posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Recurrent Implantation Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Endometrial scratch group (Active Comparator): endometrial scratch controlled ovarian hyperstimulation
  Interventions: Procedure: endometrial scratch; Procedure: controlled ovarian hyperstimulation
- Assisted hatching group (Active Comparator): assisted hatching controlled ovarian hyperstimulation
  Interventions: Procedure: assisted hatching; Procedure: controlled ovarian hyperstimulation
- ovarian stimulation only group (Sham Comparator): controlled ovarian hyperstimulation
  Interventions: Procedure: controlled ovarian hyperstimulation

INTERVENTIONS:
Procedure: endometrial scratch — midluteal endometrial scratch using Novak curette under general anesthesia in the cycle preceding stimulation
  Other Names: endometrial injury
  Arms: Endometrial scratch group
Procedure: assisted hatching — using Octax laser 20120644-laser 5452
  Other Names: laser hatching
  Arms: Assisted hatching group
Procedure: controlled ovarian hyperstimulation — using merional&/ or fostimon doses individualized as judged by patient age & ovarian reserve & monitored by follicular size & serum estradiol

SUMMARY:
300 recurrent implantation failure patients will be alternatively assigned to assisted hatching , endometrial scratch , and no treatment ,100 patients in each group

DETAILED DESCRIPTION:
Group 1 consists of 100 patients will undergo endometrial scratch followed by controlled ovarian hyperstimulation Group 2 consists of 100 patients will undergo controlled ovarian hyperstimulation& assisted hatching Group 3 consists of 100 patients will undergo controlled ovarian hyperstimulation

ELIGIBILITY:
Inclusion Criteria:

* recurrent implantation failure
* normal uterine cavity by transvaginal ultrasound

Exclusion Criteria:

* endometrial polyp or fibroid distorting the endometrium
* hydrosalpinx
* preimplantation genetic diagnosis
* severe male factor

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
number of patients with positive pregnancy test | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: suzy abdelaziz, lecturer, Principal Investigator — kasrelaini hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lacey L, Hassan S, Franik S, Seif MW, Akhtar MA. Assisted hatching on assisted conception (in vitro fertilisation (IVF) and intracytoplasmic sperm injection (ICSI)). Cochrane Database Syst Rev. 2021 Mar 17;3(3):CD001894. doi: 10.1002/14651858.CD001894.pub6. PMID 33730422